CLINICAL TRIAL: NCT05755386
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Iptacopan (LNP023) in Idiopathic Immune-complex-mediated Membranoproliferative Glomerulonephritis (IC-MPGN)
Brief Title: Study of Efficacy and Safety of Iptacopan in Participants With IC-MPGN
Acronym: APPARENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNP023B12302; 2022-002328-11 (EudraCT Number)
Expanded Access: NCT05222412 (Available)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: IC-MPGN
Keywords: LNP023; IC-MPGN; iptacopan; UPCR; eGFR; proteinuria
MeSH Terms: conditions — Proteinuria | interventions — iptacopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iptacopan 200mg b.i.d (Experimental): iptacopan 200mg b.i.d
  Interventions: Drug: iptacopan
- Placebo to iptacopan 200mg b.i.d. (Placebo Comparator): Placebo to iptacopan 200mg b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to iptacopan 200mg b.i.d. (Adults 200mg b.i.d; Adolescents 2x 100mg b.i.d)
  Arms: Placebo to iptacopan 200mg b.i.d.
Drug: iptacopan — iptacopan 200 mg b.i.d. (Adults 200mg b.i.d; Adolescents 2x 100mg b.i.d)
  Arms: iptacopan 200mg b.i.d

SUMMARY:
This study is designed as a multicenter, randomized, double-blind, parallel group, placebo-controlled study to evaluate the efficacy and safety of iptacopan (LNP023) in idiopathic immune complex mediated membranoproliferative glomerulonephritis.

DETAILED DESCRIPTION:
The purpose of this Phase III study is to evaluate the efficacy and safety of iptacopan compared to placebo (both administered in combination with standard of care) in participants (adults and adolescents aged 12-17 years) with idiopathic IC-MPGN. The study aims to demonstrate a reduction in proteinuria and improvement in estimated glomerular filtration rate (eGFR) in participants treated with iptacopan compared to placebo. Change in patient-reported fatigue will also be evaluated. Alternative complement pathway (AP) dysregulation is believed to underlie the clinical manifestations and progression of IC-MPGN. Upon completion of study treatment, participants will have the option to discontinue iptacopan treatment and enter a 30 day safety follow-up or continue iptacopan treatment by transitioning to an open label extension study (CLNP023B12001B; NCT03955445) and continue iptacopan treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients including adults (aged at least 18 years to ≤ 60 years) and adolescents (12 -17 years in non-EU countries at screening and 16-17 years in EU countries at screening).
* Diagnosis of idiopathic IC-MPGN as confirmed by kidney biopsy within 12 months prior to screening in adults and within 3 years of screening in adolescents (a biopsy report, review and confirmation by the Investigator is required). If such a biopsy is not available in an adult participant, this must be obtained at screening (performed and assessed locally for adults only).
* Prior to randomization, all participants must have been on a maximally recommended or tolerated dose of renin angiotensin system inhibitors (RASi), e.g an ACEi or ARB for at least 90 days (or as according to local guidelines). The doses of other drugs administered to reduce proteinuria and control the disease including mycophenolic acids (MPAs - mycophenolate mofetil or mycophenolate sodium), corticosteroids, SGLT2 inhibitors and mineralocorticoid receptor antagonists should be stable for at least 90 days prior to randomization
* UPCR ≥ 1.0 g/g (≥ 113 mg/mmol) sampled from the first morning void urine sample at Day -75 and Day -15
* Estimated GFR (using the chronic kidney disease [CKD]-EPI formula for adult participants and modified Schwartz formula for adolescents aged 12 to 17 years) or measured GFR ≥ 30 ml/min/1.73m2 at screening and Day -15.
* Mandatory vaccination against Neisseria meningitidis and Streptococcus pneumoniae infection prior to the start of study treatment. If the participant has not been previously vaccinated, or if a booster is required, the vaccine should be given according to local regulations at least 2 weeks prior to the first administration of study treatment. If the study treatment has to start earlier than 2 weeks post vaccination, prophylactic antibiotic treatment should be initiated in accordance with local standard of care.
* If not previously vaccinated, or if a booster is required, vaccination against Haemophilus influenzae infections should be given, if available and according to local regulations, at least 2 weeks prior to the first study treatment administration.

Exclusion Criteria:

* Participants who have undergone cell or solid organ transplantation, including kidney transplantation.
* Participants diagnosed with secondary IC-MPGN including but not limited to any of the following conditions:
* Deposition of antigen-antibody immune complexes as a result of any chronic infections, including

  * Hepatitis C virus (HCV) including HCV-associated mixed cryoglobulinemia, hepatitis B virus (HBV);
  * Bacterial-endocarditis, infected ventriculo-atrial shunt, visceral abscesses, leprosy, meningococcal meningitis; chronic bacterial infections
  * Protozoa/other infections- malaria, schistosomiasis, mycoplasma, leishmaniasis, filariasis, histroplasmosis

Renal deposition of immune complexes as a result of a systemic autoimmune disease:

* Systemic lupus erythematosus (SLE)
* Sjögren syndrome
* Rheumatoid arthritis
* Mixed connective tissue disease Deposition of monoclonal immunoglobulins because of a monoclonal gammopathy due to plasma cell or B cell disorders. Monoclonal gammopathy of undetermined significance (MGUS) confirmed by the measurement of serum free light chains or other investigation as per local standard of care.

Fibrillary glomerulonephritis

* Rapidly progressive crescentic glomerulonephritis defined as a 50% decline in the eGFR within 3 months with kidney biopsy findings of glomerular crescent formation seen in at least 50% of glomeruli on the most recent biopsy.
* Kidney biopsy showing interstitial fibrosis/tubular atrophy (IF/TA) of more than 50%.
* Participants with an active systemic bacterial, viral or fungal infection within 14 days prior to study treatment administration or the presence of fever ≥ 38°C (100.4°F) within 7 days prior to study treatment administration.
* A history of recurrent invasive infections caused by encapsulated organisms, e.g., Neisseria meningitidis and Streptococcus pneumoniae.
* The use of inhibitors of complement factors (e.g., Factor B, Factor D, complement 3 (C3) inhibitors, anti-Complement 5 (C5) antibodies, C5a receptor antagonists) within 3 months or 5 half-lives prior to the Screening visit.
* The use of immunosuppressants (except MPAs), cyclophosphamide or systemic corticosteroids at a dose >7.5 mg/day (or equivalent for a similar corticosteroid medication) within 90 days of study drug administration.
* The use of MPAs is not permitted within 90 days prior to randomization in India, as per the local health authority requirement.
* Acute post-infectious glomerulonephritis at screening, based upon the opinion of the investigator.
* Body mass index (BMI) >38 kg/m2 at screening and randomization. Body weight <35 kg at screening and randomization

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2028-10-27 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Log-transformed ratio to baseline in UPCR (sampled from a 24-hour urine collection) at 6 months. | 6 months (double-blind)
  To demonstrate the superiority of iptacopan compared to placebo in reducing proteinuria at 6 months.
Log-transformed ratio to baseline in UPCR at the 18-month visit (each study treatment arm) | 18 months
  To evaluate the effect of iptacopan on proteinuria at 18 months.
Log-transformed ratio to 12-month visit in UPCR at the 18-month visit in the placebo arm. | 18 months
  To evaluate the effect of iptacopan on proteinuria at 18 months.

SECONDARY OUTCOMES:
Change from baseline in eGFR | 12 months and 18 months
  To demonstrate the superiority of iptacopan vs. placebo in improving estimated glomerular filtration rate (eGFR).
Change in eGFR from the 12-month visit to the 18- month visit of the placebo arm | 18 months
  To evaluate the effect at 18 months of iptacopan in improving eGFR
Proportion of patients achieved a composite renal endpoint | 6 and 12 months
  To demonstrate the superiority of iptacopan vs. placebo in the proportion of participant who achieved a composite renal endpoint at 6 and 12 months (each study arm).
Change from baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) score. | 12 months
  To demonstrate the superiority of iptacopan compared to placebo in improvement of patient-reported fatigue at 12 months (each study arm).
Number of participants with abnormal vital signs, ECGs and safety laboratory measurements as well as study drug discontinuation due to an AE | up to 18 months
  To evaluate the safety and tolerability of iptacopan compared to placebo, number of participants with abnormal vital signs (msDBP/msSBP/heart rate), ECGs, safety laboratory measurements and study drug discontinuation due to an AE will be collected.
  msDBP: mean sitting diastolic blood pressure msSBP: mean sitting systolic blood pressure
Number of participants with clinically significant changes in heart rate, blood pressure, echocardiography parameters in adolescent patients | up to 18 months
  To evaluate the effect of iptacopan compared to placebo, number of participants with clinically significant changes in heart rate, blood pressure (msDBP/ msSBP), echocardiography parameters in adolescent patients will be collected
Annualized total eGFR slope estimated over 12 months. | 12 months
  To demonstrate the superiority of iptacopan vs. placebo in stabilizing eGFR
Log-transformed ratio to baseline in UPCR (sampled from a 24-hour urine collection) at 12 months. | 12 months
  To demonstrate the superiority of iptacopan compared to placebo in reducing proteinuria at 12 months of treatment.
Proportion of participants who achieved the composite renal endpoint at 18 months | 18 months
  To evaluate the effect of iptacopan on proteinuria at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (109):
- United States (16):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Univ Cali Irvine ALS Neuromuscular, Orange, California
  - UCSF, San Francisco, California
  - Olive View UCLA Medical Center, Sylmar, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Nicklaus Childrens Hospital, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Univ School of Medicine, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Col Uni Med Center New York Presby, New York, New York
  - Univ of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Prolato Clinical Research Center, Houston, Texas
  - Baylor Scott and White Research, Temple, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Santa Fe
- Brazil (12):
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Niterói, Rio de Janeiro
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Botucatu, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Canada (3):
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Aarhus N, Denmark
- France (5):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
- Germany (10):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Ulm
- Greece (6):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Heraklion Crete.
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- India (5):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (7):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Ranica, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Japan (4):
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Groningen, Netherlands
- Poland (6):
  - Novartis Investigative Site, Poznan, Greater Poland Voivodeship
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Slovakia (2):
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Košice
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Almería
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Kaohsiung City, Taiwan
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Izmir, Karsiyaka
  - Novartis Investigative Site, Köseköy, Kocaeli
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Mersin, Yenisehir
- United Kingdom (5):
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Salford
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: WCN24-1146 SAFETY AND EFFICACY OF IPTACOPAN IN ADOLESCENT PATIENTS WITH IC-MPGN in Elsivier Journal — https://doi.org/10.1016/j.ekir.2024.02.240